CLINICAL TRIAL: NCT06136195
Title: Influence of Mavoglurant on Alcohol Craving and Drinking in Heavy Drinkers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000029675; 2P50AA012870-21 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Consumption; Heavy Drinker; Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication; Alcoholism | interventions — mavoglurant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mavoglurant 1st / Placebo 2nd (Experimental): Participants randomized to the Mavoglurant 1st Arm will take a single dose of 200mg mavoglurant in the morning, prior to their 1st lab session. Then after a 5-8 day washout period, participants will have their 2nd lab session where they will take a matching placebo in the morning prior to the 2nd lab session.
  Interventions: Drug: Mavoglurant
- Placebo 1st / Mavoglurant 2nd (Experimental): Participants randomized to the Placebo 1st Arm will take a matching placebo in the morning, prior to their 1st lab session. Then after a 5-8 day washout period, participants will have their 2nd lab session where they will take a single dose of 200mg mavoglurant in the morning, prior to their 2nd lab session.
  Interventions: Drug: Mavoglurant

INTERVENTIONS:
Drug: Mavoglurant — The 200mg mavoglurant will be administered in the form of two 100mg oral tablets. Placebo will be administered with matching tablets.
  Other Names: STP7

SUMMARY:
The purpose of this research study is to find out about the effects of a drug called mavoglurant on alcohol consumption.

DETAILED DESCRIPTION:
This project will use a double-blind, placebo-controlled, within-subject design to examine mavoglurant effects on alcohol craving, drinking, and subjective responses. Non-treatment seeking, heavy drinkers with Alcohol Use Disorder (AUD) will undergo 2 lab sessions, which include a Cue Exposure (craving) Paradigm (CEP) and an Alcohol Drinking Paradigm (ADP), as well as 1-week and 1-month follow up appointments. Prior to the first lab session, participants will be randomized to receive either 200 mg of mavoglurant or placebo. For the second lab session, participants will receive the other condition, mavoglurant or placebo, that they did not receive in the first lab session. Each session will be separated by at least a 5-8 day washout period to allow for complete washout of mavoglurant. This is followed by 1-week and 1-month follow up appointments.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-50 (The lower limit is to avoid offering alcohol to individuals below the drinking age of 21. The upper age is determined by experience recruiting for our prior studies).
2. Ability to read English at 6th grade level or higher.
3. Meet DSM-V criteria for moderate or severe Alcohol Use Disorder (AUD).
4. Average weekly alcohol consumption of 30-70 standard drinks for men and 20-65 drinks for women. The lower limits are consistent with the lower sex-specific cut-offs defining high-risk drinking based on World Health Organization Risk Levels (WHO, 2000); the upper limits are designed to avoid recruiting participants whose drinking is likely to exceed the number of drinks available in the Alcohol Drinking Paradigm (ADP).

Exclusion Criteria:

1. Individuals who are seeking alcohol treatment or have been in alcohol treatment within the past 6 months.
2. Meet current Diagnostic and Statistical Manual v.5 (DSM-V) criteria for substance use disorder, except for tobacco use disorder or mild cannabis use disorder.
3. Positive urine drug screens at more than 1 baseline appointment for opiates, cocaine, benzodiazepines and barbiturates.
4. Psychotic or other severe psychiatric disorders as determined by clinical evaluation (Structured Clinical Interview for DSM-V; SCID). Note that if a subject endorses any harm/risk behaviors (e.g. suicidal/homicidal risk) a licensed clinician will be consulted immediately.
5. Regular use of psychoactive drugs, except for individuals on a stable dose of an antidepressant for at least 2 months.
6. Medical conditions that would contraindicate the consumption of alcohol or use of mavoglurant.
7. Clinically significant abnormalities in screening laboratories, including aspartate aminotransferase (AST) >3 times upper limit of normal (ULN); alanine aminotransferase (ALT) > 3 times ULN; total bilirubin >1.5 times ULN; serum creatinine >2.0 times ULN.
8. Neurological trauma or disease, delirium or hallucinations, or clinically significant or unstable medical conditions, including uncontrolled hypertension or diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic diseases, which in the opinion of the study physician and Principal Investigator, may put the patient at risk because of participation in the study.
9. Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scores of 8 or greater or a history of significant repeated alcohol withdrawals to reduce the likelihood of withdrawal symptomatology if subjects reduce their drinking.
10. Women who are pregnant or nursing.
11. Participants who refuse to use a reliable method of birth control.
12. Subjects who report disliking spirits will be excluded because hard liquor will be provided during the ADP.
13. Subjects who have taken any investigational drug within 4 weeks of the anticipated date of the first study dose.
14. Individuals who report heavy drinking days in the 2 days prior to their intake appointment but have a negative ethyl glucuronide (EtG) test to rule out subjects who are misrepresenting their drinking history.
15. Subjects who have donated blood within the past 6 weeks.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of drinks consumed | Lab Session 1 (Day 1); Lab Session 2 (5-8 days after Lab Session 1).
  The number of drinks consumed during the adlib session will be recorded
Change in craving for alcohol | Lab Session 1 (Day 1); Lab Session 2 (5-8 days after Lab Session 1).
  The Cue Exposure Paradigm (CEP) is used to measure craving for alcohol. The task uses a questionnaire that is in the form of a Visual Analog Scale (VAS). The endpoints will be marked with a 0 on the left indicating no craving and a 20 on the right indicating severe craving. Participants will indicate how strong they are craving to drink alcohol. The VAS takes 2-3 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center (SAC and SATU), New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data will be shared.